CLINICAL TRIAL: NCT01844258
Title: Modified Surgical Techniques for Pediatric Cataract Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Ophthalmologist, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCPMOH2010-China3
Record Dates: First submitted 2013-04-28; First posted 2013-05-01 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Cataract
Keywords: pediatric cataract; lens regeneration; endogenous lens epithelial stem cells; visual axis opacification; visual function
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified technique for I/A group (Experimental): * In the modified cataract surgery procedure, the size of the capsulorhexis opening will be decreased to 1.0-1.5 mm in diameter.
  * The capsulorhexis will be located in the peripheral area of the lens instead of the central area.
  * A 0.9 mm phacoemulsification probe will be used to remove the cataractous lens.
  * One drop of 0.5% or 1% atropine and an antibiotic/steroid ointment will be placed in the eye, which will then be patched.
  Interventions: Procedure: Modified technique
- Traditional technique for I/A group (Active Comparator): • In traditional technique group, the cataractous lens will be removed through an anterior continuous curvilinear capsulorhexis (ACCC) that is about 5-6 mm in diameter.
  Interventions: Procedure: Traditional technique

INTERVENTIONS:
Procedure: Modified technique — Peripheral 1-1.5 mm curvilinear capsulorhexis of anterior capsule
  Arms: Modified technique for I/A group
Procedure: Traditional technique — Central 5-6 mm curvilinear capsulorhexis of anterior capsule
  Arms: Traditional technique for I/A group

SUMMARY:
Pediatric cataract is totally different from adult cataract. There is traditionally no difference in technique between pediatric and adult cataract surgery. Opacification of the visual axis was the most frequent complication after pediatric surgery. In this clinical study, the investigators aimed to evaluate the safety and postoperative recovery of a modified technique for pediatric cataract surgery.

DETAILED DESCRIPTION:
This study is a randomized, controlled clinical trial with the following objectives:

* To determine whether infants with congenital cataract have improved visual outcomes following cataract extraction surgery using (1) the traditional capsulorhexis method or (2) our new minimally invasive method.
* To determine the occurrence of postoperative complications among infants with congenital cataract following cataract extraction surgery using (1) the traditional capsulorhexis method or (2) our new minimally invasive method.

The study is conducted for the following reasons:

* Transplantation of pluripotent stem cells represents an appealing therapeutic strategy in regenerative medicine, but its clinical applications have been hindered in part by concerns about tumorigenicity and immune rejection. The use of endogenous stem cells provides a possible solution to this problem.
* Lens regeneration has been reported in lower vertebrate animals. Furthermore, residual endogenous lens epithelial stem cells (LESCs) after lens removal in rabbits have been shown to proliferate and generate lens fibers.
* Cataract, or opacification of the lens, is a major cause of blindness worldwide. Surgery for congenital cataract carries a significant risk of complications and often requires additional surgical procedures to maintain the transparency of the visual axis.
* Implantation of intraocular lenses (IOLs) following cataract extraction is becoming increasingly common in the pediatric population. However, their use is controversial in children younger than two years old (especially not recommended in children younger than 6 months old due to the high incidences of IOL-related complications), as the refractive power of the eye continues to develop. In addition, IOLs have many limitations, including dislocation, less than ideal biocompatibility, inadequate accommodative properties, and suboptimal visual outcomes.
* The trial will demonstrate whether a modified cataract surgical technique can regenerate the lens from endogenous stem cells. It will also compare the incidence of complications and characterize visual outcomes in pediatric patients treated with the modified surgical technique versus the traditional surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month and 24 months
* Uncomplicated congenital cataract (≥ 3 mm central dense opacity) in one or both eyes with an intact non-fibrotic capsular bag
* Informed consent signed by a parent or legal guardian

Exclusion Criteria:

* Intraocular pressure >21 mmHg
* Preterm birth (<28 weeks)
* Presence of other ocular diseases (keratitis, keratoleukoma, aniridia, glaucoma) or systemic disease (congenital heart disease, ischemic encephalopathy)
* History of ocular diseases (any congenital eye diseases, such as, congenital cataract, congenital glaucoma, congenital aniridia) in the family
* History of ocular trauma
* Microcornea
* Persistent hyperplastic primary vitreous
* Rubella
* Lowe syndrome

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Incidence of opacification of the visual axis | six months

SECONDARY OUTCOMES:
Visual function in eyes treated for cataract | 6 months

OTHER OUTCOMES:
Postoperative complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center,Sun Yat-sen U, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Wilson ME Jr, Hafez GA, Trivedi RH. Secondary in-the-bag intraocular lens implantation in children who have been aphakic since early infancy. J AAPOS. 2011 Apr;15(2):162-6. doi: 10.1016/j.jaapos.2010.12.008. Epub 2011 Apr 3. PMID 21463960
- [Background] Grewal DS, Basti S. Modified technique for removal of Soemmerring ring and in-the-bag secondary intraocular lens placement in aphakic eyes. J Cataract Refract Surg. 2012 May;38(5):739-42. doi: 10.1016/j.jcrs.2012.02.023. PMID 22520301
- [Background] Shrestha UD. Cataract surgery in children: controversies and practices. Nepal J Ophthalmol. 2012 Jan-Jun;4(1):138-49. doi: 10.3126/nepjoph.v4i1.5866. PMID 22344012
- [Background] Tassignon MJ, Gobin L, Mathysen D, Van Looveren J, De Groot V. Clinical outcomes of cataract surgery after bag-in-the-lens intraocular lens implantation following ISO standard 11979-7:2006. J Cataract Refract Surg. 2011 Dec;37(12):2120-9. doi: 10.1016/j.jcrs.2011.06.025. PMID 22108108
- [Background] Amon M. Surgical management challenges and clinical results of bimanual micro-incision phacoemulsification cataract surgery in children with congenital cataract. Nepal J Ophthalmol. 2011 Jan-Jun;3(1):3-8. doi: 10.3126/nepjoph.v3i1.4270. PMID 21505539
- [Background] Nihalani BR, VanderVeen DK. Technological advances in pediatric cataract surgery. Semin Ophthalmol. 2010 Sep-Nov;25(5-6):271-4. doi: 10.3109/08820538.2010.518836. PMID 21091011
- [Background] Lin H, Chen W, Luo L, Congdon N, Zhang X, Zhong X, Liu Z, Chen W, Wu C, Zheng D, Deng D, Ye S, Lin Z, Zou X, Liu Y. Effectiveness of a short message reminder in increasing compliance with pediatric cataract treatment: a randomized trial. Ophthalmology. 2012 Dec;119(12):2463-70. doi: 10.1016/j.ophtha.2012.06.046. Epub 2012 Aug 24. PMID 22921386
- [Background] Luo L, Lin H, Chen W, Wang C, Zhang X, Tang X, Liu J, Congdon N, Chen J, Lin Z, Liu Y. In-the-bag intraocular lens placement via secondary capsulorhexis with radiofrequency diathermy in pediatric aphakic eyes. PLoS One. 2013 Apr 24;8(4):e62381. doi: 10.1371/journal.pone.0062381. Print 2013. PMID 23638058
- See also: Home page for Zhongshan Ophthalmic Center — http://www.gzzoc.com
- See also: Website for children cataract home — http://www.cnccclub.com